CLINICAL TRIAL: NCT05419362
Title: A Phase II Study to Evaluate the Safety and the Efficacy of GEN-001 in Combination With Avelumab for Patients With PD-L1 Positive Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: GEN-001 in Combination With Avelumab for Patients With PD-L1 Positive Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genome & Company (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [GNC] GEN001-201
Record Dates: First submitted 2022-06-13; First posted 2022-06-15 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GEN-001 with avelumab (Experimental): 42 patients in total with metastatic GC/Gastroesophageal Junction Adenocarcinoma who have progressed after 2 prior systemic treatments and confirmed PD-L1 positive expression will be enrolled in this study.
  Interventions: Drug: GEN-001; Drug: Avelumab

INTERVENTIONS:
Drug: GEN-001 — The capsules taken by mouth once a daily. Each capsule will contain ≥ 3x10^11 colony-forming units (CFU)
Drug: Avelumab — 800 mg given by intravenous (IV) infusion once every 2 weeks
  Other Names: Bavencio

SUMMARY:
This is a phase II, multicenter, open-label study to evaluate the antitumor activity, efficacy and safety of GEN-001 in combination with avelumab as a third line (3L) or greater line treatment which is not received the Standard of Care (SOC) for patients with PD-L1 positive advanced GC/Gastroesophageal Junction Adenocarcinoma who are not received cancer immunotherapy regimens as mono or combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable, recurrent, locally advanced or metastatic GC/Gastroesophageal Junction Adenocarcinoma
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Have adequate organ functions as defined in the protocol
* Negative childbearing potential
* Have experienced documented objective radiographic or clinical disease progression after 2 or above previous lines of standard therapy.
* PD-L1 positive
* Measurable disease as per RECIST v1.1 defined as at least 1 lesion
* Estimated life expectancy of at least 3 months
* Have ability to swallow and retain oral medication and no clinically significant gastrointestinal abnormalities

Exclusion Criteria:

* Previously received T-cell coregulatory protein inhibitors
* Has clinically significant evidence of ascites by physical exam
* Known prior severe hypersensitivity reactions to monoclonal antibodies or any component in their formulation
* Has active autoimmune disease that has required systemic treatment in the past 2 years
* Current use of immunosuppressive medication
* Have an active infection requiring antibiotics, antifungal or antiviral agents or have received a course of antibiotics within 4 weeks
* Has received a live vaccine within 4 weeks
* Known history or any evidence of active for non-infectious pneumonitis
* Prior solid organ or allogeneic stem cell transplantation
* Has had any investigational or anti-tumor treatment within 4 weeks or 5 half-life periods of starting study treatment, had any major surgeries within 4 weeks
* Has received proton pump inhibitors (PPIs) within 2 weeks
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has clinically significant (i.e., active) cardiovascular disease
* Has other persisting toxicities
* Has other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, or psychiatric conditions

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
To assess the anti-tumor activity of GEN-001, when administered as combined with avelumab | 1 years
  Objective Response (OR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Incidence of Adverse Events | 1 years
  Assessed as per CTCAE v5.0
Incidence of Laboratory abnormalities | 1 years
  Assessed as per CTCAE v5.0
Duration of response (DoR) | 1 years
  Assessed according to RECIST v1.1
Progression-free Survival (PFS) | 1 years
  Assessed according to RECIST v1.1
Overall Survival (OS) | 1 years

OTHER OUTCOMES:
Microbiota | 1 years
  fecal samples will be collected for analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jeeyun Lee, Principal Investigator — Samsung Medical Center
Locations (5):
- South Korea (5):
  - Ajou University Hospital, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No